CLINICAL TRIAL: NCT02469948
Title: Botulinim Toxin Type A Injections by Different Guidance in Stroke Patients With Spasticity on Lower Extremities
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMRPG8BC0781
Record Dates: First submitted 2015-04-15; First posted 2015-06-12 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-09

CONDITIONS: Cerebrovascular Accident
Keywords: spasticity; botulinum toxin; ultrasonography guidance; electric stimulation guidance; stroke
MeSH Terms: conditions — Stroke; Muscle Spasticity | interventions — Botulinum Toxins, Type A; Botulinum Toxins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasonography direct-guidance (Experimental): To inject Botulinum toxin type A on the spasticity lower extremity for stroke patients by Ultrasonography direct-guidance.
  Interventions: Drug: Botulinum toxin type A
- Surface anatomy landmark (Active Comparator): To inject Botulinum toxin type A on the spasticity lower extremity for stroke patients by Surface anatomy landmark.
  Interventions: Drug: Botulinum toxin type A

INTERVENTIONS:
Drug: Botulinum toxin type A — To inject Botulinum toxin type A on the spasticity lower extremity for stroke patients by Ultrasonography direct-guidance, Electric stimulation and Surface anatomy landmark.
  Other Names: Botulinum toxin

SUMMARY:
Stroke may result in lower extremity spasticity, which interfere with motor voluntary function and activities of daily living. Botulinum toxin type A (BTX-A) has been shown to improve lower extremity spasticity of stroke patients. There are no researches to compare the efficiency of BTX-A injection by different guidance methods in the deep muscles of lower extremity for stroke patients. The aims of investigator's study were to compare the effectiveness of BTX-A injection by different guidance methods (palpation of anatomical landmarks, ultrasonography direct) in deep spastic muscles of lower extremity for stroke patients with varus spasticity and spastic claw toes , and to study the correlation between muscles spasticity and elastic properties by the sonoelastography/acoustic radiation force impulse imaging and follow the change of elastic properties in spastic muscles after BTX-A injection. We will enroll 80 hemiplegic stroke patients with varus spasticity / spastic claw toes and duration more than 6 months. Under different guidance methods (palpation of anatomical landmarks, electric stimulation, ultrasonography direct and indirect methods), BTX-A will be injected to the flexor digitorum longus and posterior tibialis muscles. If the patients have moderate hallucis spasticity, flexor hallucis longus muscle will be injected. The BTX-A dose is 50 units for each muscle. Outcome measures include Modified Ashworth Scale, Brunnstrom stage, muscle power, range of motion, the visual analog scale of pain, Stroke Impact Scale, Barthel index and lower extremity function tests, balance test, Goal Attainment Scale, sonoelastography and acoustic radiation force impulse imaging. All the assessments will be performed before BTX-A injection and followed up at 1 months, 2 months, 3 months and 6 months after injection. After performing all the assessments, investigator will investigate the efficiency of BTX-A by different guidance methods.

DETAILED DESCRIPTION:
Stroke may result in lower extremity spasticity, which interfere with motor voluntary function and activities of daily living. Botulinum toxin type A (BTX-A) has been shown to improve lower extremity spasticity of stroke patients. There are no researches to compare the efficiency of BTX-A injection by different guidance methods in the deep muscles of lower extremity for stroke patients. The aims of investigator's study were to compare the effectiveness of BTX-A injection by different guidance methods (palpation of anatomical landmarks, electric stimulation, ultrasonography direct and indirect methods) in deep spastic muscles of lower extremity for stroke patients with varus spasticity and spastic claw toes , and to study the correlation between muscles spasticity and elastic properties by the sonoelastography/acoustic radiation force impulse imaging and follow the change of elastic properties in spastic muscles after BTX-A injection. We will enroll 80 hemiplegic stroke patients with varus spasticity / spastic claw toes and duration more than 6 months. Under different guidance methods (palpation of anatomical landmarks, electric stimulation, ultrasonography direct and indirect methods), BTX-A will be injected to the flexor digitorum longus and posterior tibialis muscles. If the patients have moderate hallucis spasticity, flexor hallucis longus muscle will be injected. The BTX-A dose is 50 units for each muscle. Outcome measures include Modified Ashworth Scale, Brunnstrom stage, muscle power, range of motion, the visual analog scale of pain, Stroke Impact Scale, Barthel index and lower extremity function tests, balance test, Goal Attainment Scale, sonoelastography and acoustic radiation force impulse imaging. All the assessments will be performed before BTX-A injection and followed up at 1 months, 2 months, 3 months and 6 months after injection. After performing all the assessments, investigator will investigate the efficiency of BTX-A by different guidance methods.

Two of arms:

1. ultrasonography direct-guidance: To inject Botulinum toxin type A on the spasticity lower extremity for stroke patients by Ultrasonography direct-guidance.
2. surface anatomy landmark: To inject Botulinum toxin type A on the spasticity lower extremity for stroke patients by surface anatomy landmark.

ELIGIBILITY:
Inclusion Criteria:

* ankle varus spasticity with spasticity claw toes
* MP joint and IP joint are above Modified Ashworth Scale 1 +
* ankle varus spasticity and spasticity claw toes during walking should reach median level
* patients feel pain or uncomfortable during walking due to spasticity claw toes.
* patients never accept botox, phenol and alcohol injections before.

Exclusion Criteria:

* contracture or deformity on lower extremity
* combine other systemic disease of neurological or skelectomuscular system
* patients accepted botox, phenol, alcohol injections and operation before.
* cognition disorder or aphasia after stroke
* Flexor Digitorum Longus, posterior tibialis and Flexor pollicis longus muscle has been significant atrophy .
* systemic infection
* under medication treatment of aminioglycoside or which can change neuromuskular transmission medicine
* ankle plantarflxeor contracture during walking above median level or the sore of Modified Ashworth Scale is above 2 at rest
* allergy to botox

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Modified Ashworth scale | patients will be evaluated at 4 weeks, 8 weeks, 12 weeks, 24 weeks and 1 year after injection

SECONDARY OUTCOMES:
activities of daily living | patients will be evaluated at 4 weeks, 8 weeks, 12 weeks, 24 weeks and 1 year after injection
Berg Balance Test | patients will be evaluated at 4 weeks, 8 weeks, 12 weeks, 24 weeks and 1 year after injection
Tinetti Gait Analysis | patients will be evaluated at 4 weeks, 8 weeks, 12 weeks, 24 weeks and 1 year after injection
Mini-Mental State Examination | patients will be evaluated at 4 weeks, 8 weeks, 12 weeks, 24 weeks and 1 year after injection
Stroke Impact Scale | patients will be evaluated at 4 weeks, 8 weeks, 12 weeks, 24 weeks and 1 year after injection
Fugl-Meyer Assessment Score | patients will be evaluated at 4 weeks, 8 weeks, 12 weeks, 24 weeks and 1 year after injection
Functional Ambulation Classification | patients will be evaluated at 4 weeks, 8 weeks, 12 weeks, 24 weeks and 1 year after injection

CONTACTS AND LOCATIONS:
Overall Officials: Pong Ya-Ping, MD, Study Chair — Rehabilitation
Locations (1):
- Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Stoquart GG, Detrembleur C, Palumbo S, Deltombe T, Lejeune TM. Effect of botulinum toxin injection in the rectus femoris on stiff-knee gait in people with stroke: a prospective observational study. Arch Phys Med Rehabil. 2008 Jan;89(1):56-61. doi: 10.1016/j.apmr.2007.08.131. PMID 18164331
- [Background] Caty GD, Detrembleur C, Bleyenheuft C, Deltombe T, Lejeune TM. Effect of simultaneous botulinum toxin injections into several muscles on impairment, activity, participation, and quality of life among stroke patients presenting with a stiff knee gait. Stroke. 2008 Oct;39(10):2803-8. doi: 10.1161/STROKEAHA.108.516153. Epub 2008 Jul 17. PMID 18635841
- [Background] Wissel J, Ward AB, Erztgaard P, Bensmail D, Hecht MJ, Lejeune TM, Schnider P, Altavista MC, Cavazza S, Deltombe T, Duarte E, Geurts AC, Gracies JM, Haboubi NH, Juan FJ, Kasch H, Katterer C, Kirazli Y, Manganotti P, Parman Y, Paternostro-Sluga T, Petropoulou K, Prempeh R, Rousseaux M, Slawek J, Tieranta N. European consensus table on the use of botulinum toxin type A in adult spasticity. J Rehabil Med. 2009 Jan;41(1):13-25. doi: 10.2340/16501977-0303. PMID 19197564
- [Background] Chin TY, Nattrass GR, Selber P, Graham HK. Accuracy of intramuscular injection of botulinum toxin A in juvenile cerebral palsy: a comparison between manual needle placement and placement guided by electrical stimulation. J Pediatr Orthop. 2005 May-Jun;25(3):286-91. doi: 10.1097/01.bpo.0000150819.72608.86. PMID 15832139
- [Background] Molloy FM, Shill HA, Kaelin-Lang A, Karp BI. Accuracy of muscle localization without EMG: implications for treatment of limb dystonia. Neurology. 2002 Mar 12;58(5):805-7. doi: 10.1212/wnl.58.5.805. PMID 11889247
- [Background] Yang EJ, Rha DW, Yoo JK, Park ES. Accuracy of manual needle placement for gastrocnemius muscle in children with cerebral palsy checked against ultrasonography. Arch Phys Med Rehabil. 2009 May;90(5):741-4. doi: 10.1016/j.apmr.2008.10.025. PMID 19406292
- [Background] O'Brien CF. Injection techniques for botulinum toxin using electromyography and electrical stimulation. Muscle Nerve Suppl. 1997;6:S176-80. PMID 9826989
- [Background] Berweck S, Schroeder AS, Fietzek UM, Heinen F. Sonography-guided injection of botulinum toxin in children with cerebral palsy. Lancet. 2004 Jan 17;363(9404):249-50. doi: 10.1016/S0140-6736(03)15351-2. No abstract available. PMID 14738817
- [Background] Schroeder AS, Berweck S, Lee SH, Heinen F. Botulinum toxin treatment of children with cerebral palsy - a short review of different injection techniques. Neurotox Res. 2006 Apr;9(2-3):189-96. doi: 10.1007/BF03033938. PMID 16785117
- [Background] Picelli A, Bonetti P, Fontana C, Barausse M, Dambruoso F, Gajofatto F, Tamburin S, Girardi P, Gimigliano R, Smania N. Accuracy of botulinum toxin type A injection into the gastrocnemius muscle of adults with spastic equinus: manual needle placement and electrical stimulation guidance compared using ultrasonography. J Rehabil Med. 2012 May;44(5):450-2. doi: 10.2340/16501977-0970. PMID 22549655
- [Background] Picelli A, Tamburin S, Bonetti P, Fontana C, Barausse M, Dambruoso F, Gajofatto F, Santilli V, Smania N. Botulinum toxin type A injection into the gastrocnemius muscle for spastic equinus in adults with stroke: a randomized controlled trial comparing manual needle placement, electrical stimulation and ultrasonography-guided injection techniques. Am J Phys Med Rehabil. 2012 Nov;91(11):957-64. doi: 10.1097/PHM.0b013e318269d7f3. PMID 23085706
- [Background] Lim EC, Ong BK, Seet RC. Botulinum toxin-A injections for spastic toe clawing. Parkinsonism Relat Disord. 2006 Jan;12(1):43-7. doi: 10.1016/j.parkreldis.2005.06.008. Epub 2005 Sep 29. PMID 16198612
- [Background] Suputtitada A. Local botulinum toxin type A injections in the treatment of spastic toes. Am J Phys Med Rehabil. 2002 Oct;81(10):770-5. doi: 10.1097/00002060-200210000-00009. PMID 12362118